CLINICAL TRIAL: NCT03745339
Title: Outcome Inference in the Sensory Preconditioning Task in Opioid-use Disorder
Status: Recruiting | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919019; 19-DA-N019
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01-05

CONDITIONS: Opioid-Related Disorders; Drug Addiction
Keywords: Addiction; Orbitofrontal Cortex; Associative Learning; Implicit Learning; Natural History
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Abstinent OUD: Men and women with history of OUD, but abstinent for at least 3 weeks and not in agonist treatment
- Controls: Men and women with no history of a substance-use disorder (except nicotine, for matching purposes) and not using any drug for nonmedical purposes
- In-treatment OUD: Men and women with opioid use disorder (OUD) being treated with an agonist (buprenorphine or methadone)

SUMMARY:
Background:

People with addictions often find it hard to choose the long-term benefits of abstinence over the short-term effects of using drugs. Researchers think this is partly due to parts of the brain involved in certain types of learning and decision-making. Researchers want to test these basic functions using a simple task with pictures and odors.

Objective:

To see if performance in a learning task differs between people who have opioid-use disorder and people who don t.

Eligibility:

Adults 21-60 years old who are willing to fast for at least 6 hours and smell food odors. Those with an opioid-use disorder must either not use for at least 3 weeks or be in treatment.

Design:

Participants will have 1 visit that will take up to 5 hours.

Before the visit, participants will be asked to not eat or drink anything except water for at least 6 hours.

At the visit, participants will be checked for signs of intoxication.

Participants will give urine and breath samples.

Participants will have tests of learning and behavior. They will look at shapes on a computer screen. The shapes will be paired with different food odors.

The odors will come from a sterile tube placed under the nose.

Participants will have their breathing monitored with a belt around the upper abdomen.

About 30 days and 60 days later, participants will be called and asked about their drug use over the past 30 days.

DETAILED DESCRIPTION:
Background. People with substance-use disorders may have difficulty guiding their behavior on the basis of not-yet-experienced outcomes such as long-term effects of substance use. Use of mental inferences about future outcomes can be tested in a relatively simple laboratory task called sensory preconditioning.

Objective. To test whether sensory-preconditioning performance is worse in people with opioid use disorder (OUD) than in healthy, demographically matched controls. To increase generalizability, we will examine OUD participants who are in agonist treatment (abstinent or not) and OUD participants who are abstinent but not in treatment. We do not have a hypothesis about differences between those two groups, but we hypothesize that among agonist-treated OUD participants, performance will correlate with degree of abstinence.

Participant population. We will enroll 3 groups of men and women: (1) history of OUD, but abstinent for at least 3 weeks and not in agonist treatment, (2) OUD being treated with an agonist (buprenorphine or methadone), (3) no history of a substance-use disorder (except nicotine, for matching purposes) and not using any drug for nonmedical purposes.

Experimental design. Between-groups cross-sectional single-session laboratory study, with telephone follow-up at 30 and 60 days.

Methods. Each participant will participate in a sensory preconditioning task conducted in a single session. The task uses food odors delivered via nasal cannula and paired with visual cues on a computer screen. There are three phases: (1) Preconditioning, in which 2 pairs of visual cues (A+B, C+D) are shown on the computer screen; participants should acquire automatic associations between A+B and between C+D. (2) Conditioning, in which participants learn associations between the second cue of each pair (B and D) and either a sweet odor (B1), a savory odor (B2), or no odor (D); and (3) Probe Test, in which participants predict whether a visual cue will be paired with the sweet odor, the savory odor, or no odor, by pressing a left, middle, or right button. No odors are actually delivered in the probe test. The test of inference-guided behavior is the ability to associate visual cues A and C with an odor despite their never having been directly paired with an odor. In telephone follow-up at 30 and 60 days, participants will be asked to report drug use and associated problems since the session or follow-up call.

Primary outcome measures. (1) Value-based outcome inference as measured using responding to cues A minus C in the probe test. It is defined as the percentage of trials in which behavioral responses indicate a prediction of any odorant (sweet or savory), independent of whether this prediction is correct. Responding to cues B minus D will be used as a covariate to control for differences in olfactory acuity and non-inference-based task performance.

Secondary outcome measures. (1) The percentage of trials in which the odor prediction is correct. (2) Response latency per cue type. (3) Amplitude and (4) latency of respiratory (sniff) responses per cue type. (5) Acquisition (% responding to B minus D in the last run of conditioning) during the training portion of the inferencing task. (6) Drug use and associated problems at follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA:

The enrollment target for the protocol is 120 (40 healthy controls, 40 patients on agonist maintenance, and 40 participants who have met DSM 5 criteria for OUD, but are now abstinent (for at least 3 weeks) and not on agonist maintenance.

All Participants

* Age between 21 and 65 years inclusive. Rationale: objective olfactory impairment grows more prevalent with age; after age 53, the prevalence is 24.5%, increasing to 62.5 % in people aged 80-97 years.
* Willing to fast for at least 6 hours prior to the study session and be exposed to food odors. These will be assessed with the "019 Additional History Form" questionnaire.

Additional Criteria for Abstinent OUD group

* History of opioid-use disorder (DSM-5), to be assessed via the Mini International Neuropsychiatric Interview (MINI) or the Structured Clinical Interview for DSM-5 (SCID). History of SUDs can include substances in addition to opioids (e.g., cocaine).
* Abstinent > 3 weeks from all illicit substances (tobacco smoking and nondependent drinking permissible), to be assessed via 30-day timeline follow-back calendar. (Current abstinence will be confirmed via urine screen: see exclusion criteria.) Rationale: Although heterogeneity will be considerable, what all enrollees will have in common is having become abstinent from opioids long enough to be past withdrawal symptoms. Their heterogeneity in duration of abstinence and other drug-history measures will enable us to examine relationships between those things and inferencing performance.

Additional Criteria for In-treatment OUD group

-Current enrollment in treatment for OUD with buprenorphine or methadone (>3 weeks on stable dose). Current use of illicit substances during treatment is permissible but not required. Rationale: Again, heterogeneity will be considerable, but what all enrollees will have in common is having sought treatment for their OUD and being currently maintained on an agonist that permits adaptive everyday functioning. Their heterogeneity in ongoing use of illicit substances will enable us to examine relationships between inferencing performance and treatment response.

EXCLUSION CRITERIA:

All participants

* Anosmia, dysosmia, or hyposmia (poor olfactory function), to be assessed via Sniffin Sticks threshold test <4 or via Sniffin Sticks odor identification test <10.
* History of any neurological condition resulting in inability to perform study task. Examples include but not limited to degenerative processes of the CNS (Parkinson disease, Alzheimer disease); other neurologic diseases (Huntington disease, multiple sclerosis, other motor-neuron diseases); inflammatory conditions (sarcoidosis, Wegener granulomatosis); or significant cerebrovascular disease including (but not limited to) epilepsy, stroke, or meningitis; traumatic brain injury (TBI) or major head trauma with sustained loss of consciousness (>30 min). To be assessed by history and physical and evaluation to sign screening consent. Eligibility will be determined based on MAI review of participants ability to perform study task. MAI will consider but is not limited to H and P results for mental status exam, language exam, and attention span exam. Rationale: any of these could impair task performance.
* History of current (past 12 months) uncontrolled DSM-5 major psychiatric disorder including major affective disorder, obsessive-compulsive disorder, schizophrenia, and PTSD. (Candidates will not be excluded for a history of major psychiatric disorder that is now being successfully treated.) To be assessed by MINI or SCID interview. Rationale: could impair task performance.
* History of anaphylaxis due to, e.g., significant asthma, food or non-food allergy, or intolerance to odors (including latex, detergents, soaps, etc.). To be assessed by history and physical. Rationale: could make odorant exposure risky.
* Current use of medications or substances that affect alertness and that cannot be withheld on the morning of the study visit (e.g., barbiturates, benzodiazepines, cannabinoids, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, etc.). To be assessed by history and physical. Whether candidate will be requested to withhold any medication will be determined based on MAI judgment. Additionally, if participant has a BrAC >0.08, MAI will use clinical judgement to determine if participant should be rescheduled. Rationale: could impair task performance.
* For women: pregnancy. To be assessed by history and physical and by urine testing. Rationale: Could affect task performance-physiological and hormonal changes during pregnancy influence rhinological function.
* Any other medical illness or condition that in the judgment of the investigators is incompatible with study participation.

Additional criteria for Control Group

* History of a substance-use disorder (except nicotine, for matching purposes), or current use of any drug for nonmedical purposes. Controls, who cannot have a history of OUD, will be assessed by their medical history and physical examination for the presence of any signs or symptoms consistent with opioid withdrawal. Any Control with any sign or symptom consistent with opioid withdrawal will be evaluated by the MAI to rule out opioid withdrawal if possible.
* Urine positive for any illicit drug. Rationale: Controls should have no drug use. A UDS that is positive for a prescribed medication that the MAI has determined is not due to illicit drug use will not be exclusionary.

Additional criteria for Abstinent Group

* Urine positive for any illicit drug. Rationale: Abstinent OUD group should have no drug use in the last 3 weeks which would include the several-day time frame to which urine screens are sensitive. A UDS that is positive for a prescribed medication that the MAI has determined is not due to illicit drug use will not be exclusionary.
* Current signs or symptoms of opioid withdrawal. These will be assessed in the Abstinent group via the Clinical Opioid Withdrawal Scale (COWS) and the Subjective Opioid Withdrawal Scale (SOWS).

Additional criteria for In-treatment OUD group

-Urine negative for opioid agonist that the participant is taking as part of their OUD treatment. Rationale: In-treatment OUD group should be in treatment. A negative test suggests the participant is not adhering to their treatment plan. In-treatment OUD participants may test positive for other substances as well as their opioid agonist because they may have ongoing illicit drug use.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Outcome inferencing in the probe test | During task
  Percentage of trials with cues A and C in which the participant predicts any odor (sweet or savory), regardless of whether the prediction is correct.

SECONDARY OUTCOMES:
Percentage of trials in which the odor prediction is correct. | During task
  Task-performance measure of secondary interest
Response latency per cue type | During task
  Task-performance measure of secondary interest
Amplitude of respiratory (sniff) responses per cue type | During task
  Task-performance measure of secondary interest
Latency of respiratory (sniff) responses per cue type | During task
  Task-performance measure of secondary interest
Drug use at follow-up | 30 and 60 days
  Clinical-outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kahnt, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schoenbaum G, Chang CY, Lucantonio F, Takahashi YK. Thinking Outside the Box: Orbitofrontal Cortex, Imagination, and How We Can Treat Addiction. Neuropsychopharmacology. 2016 Dec;41(13):2966-2976. doi: 10.1038/npp.2016.147. Epub 2016 Aug 11. PMID 27510424
- [Background] Jones JL, Esber GR, McDannald MA, Gruber AJ, Hernandez A, Mirenzi A, Schoenbaum G. Orbitofrontal cortex supports behavior and learning using inferred but not cached values. Science. 2012 Nov 16;338(6109):953-6. doi: 10.1126/science.1227489. PMID 23162000
- [Background] BROGDEN WJ. Sensory pre-conditioning of human subjects. J Exp Psychol. 1947 Dec;37(6):527-39. doi: 10.1037/h0058465. No abstract available. PMID 18920626